CLINICAL TRIAL: NCT00441974
Title: A 48-week Multi-centre, Open-label, Local Phase IV Study to Demonstrate the Efficacy and Safety of Adefovir Dipivoxil Tablets (10mg) in Chinese Subjects With Compensated Chronic Hepatitis B
Brief Title: Adefovir Dipivoxil For The Treatment Of Chinese Compensated Chronic Hepatitis B(CHB)Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADF108356
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Hepatitis B
Keywords: adefovir dipivoxil; compensated; chronic hepatitis B; Chinese
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil

ARMS (1):
- Single arm adefovir dipivoxil (Experimental): adefovir dipivoxil once daily orally 10 mg
  Interventions: Drug: adefovir dipivoxil

INTERVENTIONS:
Drug: adefovir dipivoxil — adefovir dipivoxil once daily one tablet 10mg orally

SUMMARY:
This 48-week open-label study of local manufactured adefovir dipivoxil Tablet evaluates the efficacy and safety of adefovir 10mg once daily in Chinese subjects with compensated CHB. Primary endpoint is proportion of subjects achieving HBV DNA undetectable (<=1000 copies/mL by by Roche COBAS AMPLICOR HBV MONITOR Test) at week 48. Approximately 1250 patients will be recruited in 30 study centers in China. The subjects are offered 48 weeks of open label adefovir dipivoxil treatment, with assessments every three months, after with is a 12-week post study treatment follow-up prior to study completion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18-65 years inclusive
* Documented chronic hepatitis B infection determined by the presence of serum HBsAg for a least 6 months
* Serum HBV DNA ≥105 copies/ml for HBeAg positive subjects or ≥104 copies/ml for HBeAg negative subjects (Real-time PCR, LLQ=1000cp/ml) at study screening (within 2 weeks before baseline), respectively.
* ALT value ≥2 times the upper limit of normal (ULN) at the time of screening, as determined using laboratory ranges and documented ALT abnormal within 6 month prior the study screening.
* Compensated liver disease with the following laboratory and clinical parameters study screening:
* prothrombin time ≤ 2 seconds above normal direct bilirubin
* Albumin≥35g/L
* Total bilirubin ≤2.5mg/dL (≤ 43 µmol/L) or normal direct bilirubin
* No history of variceal bleeding
* No history of encephalopathy
* No history of ascites
* Willing and able to undergo two liver biopsies (prior to dosing, and after 48 weeks of therapy; only apply to subjects who are enrolled to the sites where liver biopsy is required).
* Agree not to participate in any other investigational trials or to undertake other HBV systemic antiviral regimens during participation in this study

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Any serious or active medical or psychiatric illnesses other than hepatitis B which, in the opinion of the investigator, would interfere with patient treatment, assessment or compliance with the protocol. This would include, may not limit to, renal, cardiac, pulmonary, vascular, neurogenic, digestive, metabolic (diabetes, thyroid disorders, adrenal disease), immunodeficiency disorders, active infection or cancer.
* Documented evidence of active liver disease due to other causes including
* co-infection hepatitis C (HCV), Subjects who are anti-HCV positive and in whom HCV RNA is undetectable are considered to be HCV seropositive and will not be eligible
* co-infection with hepatitis delta (HDV)
* co-infection with HIV
* autoimmune hepatitis (antinuclear antibody titre>1:160)
* Alanine aminotransferase(ALT) > 10 times ULN at screening or history of acute exacerbation leading to transient decompensation
* Serum alpha fetoprotein (AFP) >50 ng/mL.
* Hepatocellular carcinoma as evidenced by one of the following:
* suspicious foci on ultrasound or radiological examination
* where no positive ultrasound finding, but serum alpha-fetoprotein > 100ng/ml
* Adequate renal function defined as serum creatinine >1.5 mg/dL (>130 µmol/L)
* Adequate hematological function defined as:
* Absolute neutrophil count <1 x 10³/mm³ (1 x 10^9/L)
* Platelets<80 x 10³/mm³ (80 x 10^9/L); platelets<100 x 10³/mm³ (100 x 10^9/L)
* Hemoglobin<12g/dL (120 g/L)(males) or <10 g/dL (100 g/L) (females)
* Active alcohol or drug abuse or history of alcohol or drug abuse considered by the investigator to be sufficient to hinder compliance with treatment, participation in the study or interpretation of results.
* Use of immunosuppressive therapy, immunomodulatory therapy (including interferon or thymosin), systemic cytotoxic agents within the previous 6 months or during the study.
* Use of chronic anti-viral agents(e.g. lamivudine, adefovir dipivoxil, entecavir, famciclovir, tenofovir, FTC, ganciclovir, DAPD, LfMA, HBIg, etc.), Chinese herbal medicines known to have activity against HBV within the previous 3 months or during the study; use of agents with effect of ALT reduction (e.g. schisandra agents) during the study.
* Received nephrotoxic drugs (e.g., aminoglycosides, amphotericin B, vancomycin, cidofovir, foscarnet, cis-platinum, pentamidine etc.) or competitors of renal excretion (e.g., probenecid within 2 months prior to study screening or the expectation that patient will receive any of these during the course of the study.
* Received hepatotoxic drugs (e.g., anabolic steroids, ketaconazole, itraconazole, isoniazid, rifampin, rifabutin) within 2 months prior to study screening or expected to receive these during the course of the study.
* Previous (or planned) participation in an investigational trial involving administration of investigational compound within 2 months prior to the study screening.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1470 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- China (14):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Chongquin
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg Adefovir Dipivoxil: Adefovir Dipivoxil (ADV) 10 mg tablets once daily for 48 weeks
Period: Overall Study
Arm/Group | 10 mg Adefovir Dipivoxil
Started | 1470
Completed | 1342
Not Completed | 128
Not completed — Adverse Event | 6
Not completed — Consent Withdrawn | 35
Not completed — Lost to Follow-up | 80
Not completed — Protocol Violation | 7

BASELINE CHARACTERISTICS:
Arm/Group | 10 mg Adefovir Dipivoxil
Number analyzed (Participants) | 1467
Age Continuous [Mean (Standard Deviation); unit: years] — The Intent-to-Treat (ITT) Population was used as the analysis population.
  years | 31.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants] — The Intent-to-Treat (ITT) Population was used as the analysis population.
  Participants
    Female | 291
    Male | 1176
Race/Ethnicity, Customized [Number; unit: participants] — The Intent-to-Treat (ITT) Population was used as the analysis population.
  participants
    Asian | 1467

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving HBV DNA (Hepatitis B Virus Deoxyribonucleic Acid) <1000 Copies/Milliliter at Week 48
Description: HBV (Hepatitis B Virus) DNA level was tested by real-time Polymerase Chain Reaction at Week 48.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Number; unit: participants
Groups:
- HBeAg+ at Baseline: Participants who had detectable HBeAg (Hepatitis B e Antigens) as measured by a local laboratory
- HBeAg- at Baseline: Participants who had undetectable HBeAg as measured by a local laboratory
- Total: Total of HBeAg+ and HBeAg- participants
Arm/Group | HBeAg+ at Baseline | HBeAg- at Baseline | Total
Number analyzed (Participants) | 1108 | 359 | 1467
participants
  HBV DNA <1000 copies (cp)/mL | 341 | 243 | 584
  HBV DNA >1000 cp/mL | 767 | 116 | 883

2. Secondary Outcome: Number of HBeAg Positive Participants Achieving Histological Improvement at Week 48
Description: Histological improvement (defined as a ≥2 point reduction in the Knodell necroinflammation score without worsening fibrosis) was accessed by two pathologists in HBeAg-positive participants undergoing liver biopsy at baseline and week 48/withdrawal. Knodell/Histological Activity Index (HAI) score = combined scores for necrosis, inflammation, and fibrosis and is the sum of scores for periportal bridging necrosis (0-10: none=0, multilobular necrosis=10), intralobular degeneration and focal necrosis and portal inflammation (0-4: none=0, marked=4), and fibrosis (0-4: none=0, cirrhosis=4).
Time Frame: Week 48
Population: HBeAg positive chronic hepatitis B participants who underwent liver biopsy at Week 48
Measure: Number; unit: participants
Arm/Group | HBeAg+ at Baseline
Number analyzed (Participants) | 71
participants
  Histological improvement | 46
  No histological improvement | 25

3. Secondary Outcome: Ranked Assessment of Liver Histology in HBeAg Positive Participants From Baseline to Week 48
Description: A ranked assessment with the Knodell/HAI scoring system that represents the sum of scores for periportal bridging necrosis (0-10: none=0, moderate piecemeal necrosis plus bridging necrosis=5, multilobular necrosis=10); interlobular degeneration and focal necrosis (0-4: none=0, marked=4); portal inflammation (0-4: none=0, marked=4) and fibrosis (0-4: none=0, fibrous portal expansion=1, bridging fibrosis=3, cirrhosis=4) was carried out by two pathologists in the HBeAg positive participants who underwent liver biopsy at baseline and Week 48/withdrawal.
Time Frame: Baseline to Week 48
Population: HBeAg positive chronic hepatitis B participants who underwent liver biopsy at Week 48
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | HBeAg+ at Baseline
Number analyzed (Participants) | 71
points on a scale
  Knodell score at baseline | 7.7 (3.9)
  Knodell score at Week 48/withdrawal | 5.2 (2.6)
  Necroinflammation score at baseline | 6.3 (3.2)
  Necroinflammation score at Week 48/withdrawal | 3.6 (1.9)
  Fibrosis score at baseline | 1.4 (1.0)
  Fibrosis score at Week 48/withdrawal | 1.5 (0.9)

4. Secondary Outcome: Change From Screening in Median Serum HBV DNA at Weeks 24 and 48
Description: The HBV DNA level was tested in blood serum by real-time Polymerase Chain Reaction with the LLD (lower limit of detection) as 300 copies/milliliter (cp/mL) at screening, week 24, and week 48 in a central laboratory. The change in HBV DNA from screening to week 24 and week 48 was conducted.
Time Frame: Weeks 24 and 48
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Median (Full Range); unit: log10 copies/milliliter
Arm/Group | HBeAg+ at Baseline | HBeAg- at Baseline
Number analyzed (Participants) | 1108 | 359
log10 copies/milliliter
  Serum HBV DNA Change at Week 24 | -4.1 [-9.4 to 2.8] | -4.3 [-9.0 to 1.8]
  Serum HBV DNA Change at Week 48 | -4.6 [-9.4 to 3.5] | -4.6 [-9.0 to 1.6]

5. Secondary Outcome: Number of Participants Achieving ALT (Alanine Aminotransferase) Normalization at Week 48
Description: Elevated serum ALT levels are defined as serum ALT levels greater than the upper limit of the normal range (ULN), as determined using local laboratory ranges. ALT normalization was defined as ALT measurements at or below the ULN after a baseline value above the ULN.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Number; unit: participants
Arm/Group | HBeAg+ at Baseline | HBeAg- at Baseline
Number analyzed (Participants) | 1108 | 359
participants
  ALT normalization | 780 | 258
  ALT non-normalization | 328 | 101

6. Secondary Outcome: Number of HBeAg Positive Participants Achieving HBeAg Loss and HBeAg Seroconversion at Week 48
Description: HBeAg loss and HBeAg seroconversion (HBeAg loss and HBeAb detected) were assessed in participants who were HBeAg positive at Weeks 0 and 48. Confirmed HBeAg loss was defined as undetectable HBeAg.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Population: all HBeAg positive participants who actually received the study medication at least once
Measure: Number; unit: participants
Arm/Group | HBeAg+ at Baseline
Number analyzed (Participants) | 1108
participants
  HBeAg loss | 289
  HBeAg seroconversion | 151

7. Secondary Outcome: Number of Participants With ADV-associated Resistance at Week 48
Description: Week 48 serum samples from participants, who reached a HBV DNA breakthrough or have HBV DNA≥5 log copies/mL at Weeks 24 and 48 were assessed for the development of ADV (Adefovir dipivoxil) mutation (N236T and A181V) in the HBV polymerase. Virologic breakthrough was defined as an increase in the level of HBV DNA 1 log10 copy/mL from Week 24 to Week 48. ADV-associated resistance was defined as participants with both virologic breakthrough and ADV mutation.
Time Frame: Week 48
Population: Intent-to-Treat (ITT) Population: all participants who actually received the study medication at least once.
Measure: Number; unit: participants
Arm/Group | 10 mg Adefovir Dipivoxil
Number analyzed (Participants) | 1467
participants
  HBV DNA breakthrough | 66
  ADV-associated resistance | 7
  HBV DNA≥5 log copies/ml at Weeks 24 and 48 | 322

ADVERSE EVENTS:
Arm/Group | 10 mg Adefovir Dipivoxil
Serious Adverse Events (participants affected / at risk) | 18
Other Adverse Events (participants affected / at risk) | 86
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 10 mg Adefovir Dipivoxil
Hepatic mass (Hepatobiliary disorders) | 1/1467
Hepatitis B (Infections and infestations) | 7/1467
Alanine aminotransferase increased (Investigations) | 2/1467
Transaminases increased (Investigations) | 1/1467
Muscle mass (Musculoskeletal and connective tissue disorders) | 1/1467
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/1467
Nephrolithiasis (Renal and urinary disorders) | 1/1467
Breast cancer (Reproductive system and breast disorders) | 1/1467
Ovarian cyst (Reproductive system and breast disorders) | 1/1467
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 10 mg Adefovir Dipivoxil
Nasopharyngitis (Infections and infestations) | 86/1467

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.